CLINICAL TRIAL: NCT03279484
Title: Safety and Electrical Performances Evaluation of Navigo Leads Equipped With IS4 Connector
Acronym: NAVIGATOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCPL01
Record Dates: First submitted 2017-09-01; First posted 2017-09-12 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-01

CONDITIONS: Arrythmia, Implatable Cardioverter Defibrillation, Lead
Keywords: safety , electrical performance
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: NAVIGO 4LV LV leads are available as "S shaped"(NAVIGO 4LV 2D) , "U shaped" (NAVIGO 4LV ARC) and "straight"( NAVIGO 4LV Pilot) models. All the models are available in 78 cm and 88 cm long versions. All models are designed for multipolar pacing (4 electrodes) and all of them have a quadripolar IS4 connector (IS4_LLLL).
  The NAVIGO 4LV leads are steroid eluting to avoid adverse effects due to inflammation reaction of the myocardium after positioning of the lead, and therefore to limit the acute pacing threshold peak. The steroid collar design is the same as the one used in all other LIVANOVA leads
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAVIGO 4LV implant (Experimental): All patients will be attempted to implant or implanted with NAVIGO 4LV lead
  Interventions: Device: NAVIGO 4LV lead implant

INTERVENTIONS:
Device: NAVIGO 4LV lead implant — All patients will be attempted to implant or implanted with NAVIGO 4LV lead

SUMMARY:
The primary objective of this study is to assess the safety and electrical performance of Left ventricular (LV) NAVIGO 4LV leads, pre-shaped (S-shaped&U-shaped: NAVIGO 4LV 2D, NAVIGO 4LV ARC) and Straight (NAVIGO 4LV PILOT), with IS4 connector

DETAILED DESCRIPTION:
The devices under investigation, NAVIGO 4LV models Pilot, 2D , and ARC are the new quadripolar coronary venous leads with polyurethane lead body, intended to be used with defibrillators with ventricular resynchronization therapy.

The new lead design with the presence of 4 electrodes that allows several combinations in programming pacing vectors, is intended to benefit both the patients by improving response to therapy, overcoming high pacing threshold and avoiding phrenic nerve stimulation, and the investigators by reducing the number of re-interventions needed.

This clinical investigation is a pre-market release study intended to analyze safety and electrical performance of NAVIGO 4LV leads pre-shaped (S-shaped & U-shaped) and Straight leads models. The primary endpoint data will be used to support the achievement of the CE mark of NAVIGO 4LV leads.

The primary endpoints will be evaluated at 1 month post-implantation; secondary endpoints will be evaluated up to 2 years post-implantation. The duration of patient inclusion will be approximately 10 months for pre-shaped NAVIGO family (S-shaped &U-shaped) and approximately 21 months for straight ones.

The post implant follows-up visits will take place at Hospital discharge, weeks 10, 6 months and every 6 months until 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting a CRT-D indication as detailed in the ESC guidelines
* Primary implant of a PLATINIUM 4LV CRTD or upgrade from an existing ICD connected to a RV lead with a DF4 connector (DF4LLHH) to a PLATINIUM 4LV CRT-D
* Signed and dated informed consent

Exclusion Criteria:

* Patients for whom a maximum single dose of 300 µg dexamethasone sodium phosphate (DSP) eluted from the NAVIGO 4LV lead maybe contraindicated
* Venous anomalies precluding transvenous implant (contraindication of a Pacemaker or ICD implant)
* Active myocarditis, pocket and/or lead infection
* Stroke/myocardiaI infarction one month prior to implant
* Already included in another clinical study that could confound the results of this study.
* Inability to meet Follow-up visits at the implanting centre as defined in the investigational plan.
* Patient less than 18 years old or under guardianship
* Known pregnancy, women in lactation period or in childbearing age without an adequate contraceptive method (failure rate < 1%)
* Drug addiction or abuse

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Estimated)
Dates: Start 2017-11-24 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
LV lead Safety at 10 weeks | 10 weeks after implant
  Freedom from LV lead-related complications, defined as any investigational device deficiency or any serious adverse device event (SADE) that resulted in patient death or required a re-intervention (not including re-programming) that occurred within 30 days after successful implant of the CRT-D system
LV lead Performance at 10 weeks | 10 weeks after implant
  Successful performance defined as LV pacing threshold at 10 weeks < 2.5 V/0.5 ms observed on at least one pacing vector and absence of phrenic nerve stimulation at programmed pacing amplitude

SECONDARY OUTCOMES:
Electrical performance | through study completion, an average of 6 month
  LV pacing threshold amplitude (V) and LV pacing impedance (Ohm)
Rate of patients free from LV lead-related complications | through study completion, an average of 6 month
  Freedom from LV lead-related complications defined as any investigational device deficiency or any serious adverse device event (SADE) that resulted in patient death or required a re-intervention (not including re-programming)
LV lead-related SAEs | through study completion, an average of 6 month
  Serious Adverse Event LV related
Lead handing assessment of NAVIGO 4LV leads through a questionnaire | Implant
  A questionnaire on lead handling will track opinion from the investigator, comparing his assessment with this lead to device he is accustomed to implant
NAVIGO 4LV lead implant success rate on enrolled population | Enrollment
  To report the NAVIGO 4LV lead implant success rate
Number of patients with at least 2 pacing vectors with pacing threshold < 2.5 V at 0.5 ms and no phrenic nerve stimulation | 10 weeks
  To report the number of patients with at least 2 pacing vectors with pacing threshold < 2.5 V at 0.5 ms and no phrenic nerve stimulation
Number of patients with MP pacing activated | through study completion, an average of 6 month
  To report the number of patients with MP pacing activated
Rationale to activate MP | through study completion, an average of 6 month
  To report the reason why physician decide to activate MP to the patient
Number of patients with of at least one MP configuration with no phrenic nerve stimulation at programmed pacing amplitude | through study completion, an average of 6 month
  To report the number of patients with at least one MP configuration with no phrenic nerve stimulation at programmed pacing amplitude
Number of patients at each final programmed pacing vector and changes | through study completion, an average of 6 month
  To report number of patients at each final programmed pacing vector and changes

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gabriel Martinez Martinez, Principal Investigator — Hospital General Universitario Alicante Spain
Locations (38):
- France (13):
  - CHRU Brest, Brest
  - CHRU Hopital Trousseau, Chambray-lès-Tours
  - CH Robert Boulin, Libourne
  - CHU Hôpital Nord - Marseille, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - CH Annecy Genevois, Metz-Tessy
  - Groupe Hospitalier Paris St Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Bordeaux, Pessac
  - CHU Hopital Charles Nicolle, Rouen
  - CHU Rangueil, Toulouse
  - Centre Hospitalier de Valence, Valence
  - CHRU Brabois, Vandœuvre-lès-Nancy
- Germany (10):
  - Herz- und Gefässzentrum Bad Bevensen, Bad Bevensen
  - Herz- und Diabeteszentrum, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Evangelisches Krankenhaus, Bielefeld
  - Klinikum Coburg, Coburg
  - Kardiologie Darmstadt, Darmstadt
  - Universitäts-Herzzentrum Freiburg, Freiburg im Breisgau
  - Albertinen-Krankenhau, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitatsklinikum, Würzburg
- Italy (3):
  - Az. Osp-Univ. Ospedali Riuniti Umberto I-Lancisi-Salesi, Ancona
  - Ospedale Universitario Di Pisa, Pisa
  - Az. Osp. Univ. S. Maria della Misericordia, Udine
- ISALA Klinieken, Zwolle, Netherlands
- Portugal (6):
  - Centro Hospitalar Lisboa Ocidental -Hospital de Santa Cruz (CHLO), Carnaxide
  - Centro Hospitalar Universitário de Coimbra -Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar e Universitário de Coimbra - Hospital Geral, Coimbra
  - CHCL - Hospital Santa Marta, Lisbon
  - Centro H. Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto CHP Hospital de Santo Antonio, Porto
- Spain (5):
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Gregorio Marañón, Madrid
  - H. Universitario Central de Asturias, Oviedo
  - Hospital Universitario La Fe, Valencia
  - Complejo Hospitalario Universitario de Vigo - Hospital Alvaro Cunqueiro, Vigo